CLINICAL TRIAL: NCT06923358
Title: Virtual Nature as a Health-promoting Intervention for Nursing Home Residents With Dementia - a Randomized Controlled Trial
Brief Title: Virtual Nature as a Health-promoting Intervention for Nursing Home Residents With Dementia
Acronym: VR&Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South-Eastern Norway (Other)
Collaborators: Drammen municipality, Norway (Unknown)
Responsible Party: Principal Investigator, Giovanna Calogiuri, Professor, University of South-Eastern Norway
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 819127
Record Dates: First submitted 2025-03-06; First posted 2025-04-11 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dementia; Nursing Home Resident; Virtual Reality; Quality of Life; Mental Health
Keywords: Virtual nature
MeSH Terms: conditions — Dementia; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Nature intervention (VN) (Experimental): A 12-week virtual nature (VN) intervention, alongside regular medications and nursing home activities.
  Interventions: Other: Virtual Nature intervention (VN)
- Control (TAU) (No Intervention): Only the regular medications and nursing home activities ("treatment as usual")

INTERVENTIONS:
Other: Virtual Nature intervention (VN) — The intervention will consist of a 12-week virtual nature program in which participants will engage in two sessions per week. During each session, they will watch a 10-minute 360° video depicting a natural setting. Participants will select videos from a curated library of nature scenarios filmed by researchers in locations near or within the same region as their nursing homes. The videos will showcase various seasons in Norway (spring, summer, fall, and winter) and include popular activities such as hiking and cross-country skiing. The videos will be played using a Meta Quest 3 headset, with sessions conducted in participants' rooms by nursing home staff-except for the first session, which will be facilitated by the researchers.
  Arms: Virtual Nature intervention (VN)

SUMMARY:
Rationale and Objectives:

Despite significant efforts from healthcare professionals, nursing home residents with dementia often face isolation and a reduced quality of life. Increasing attention has been given to digital solutions as a complement to pharmaceutical treatments. In particular, Virtual Nature (VN; i.e., virtual reality simulations that simulate nature experiences) has emerged as a promising, cost-effective approach to enhancing quality of life and slowing cognitive decline in nursing home residents with dementia. This project aims to assess the long-term effects of a VN intervention on various health and well-being indicators in nursing home residents with dementia.

Design:

The study will be conducted as a randomized controlled trial with parallel conditions. Participants will be randomly assigned to either a treatment or a control group. The treatment group will undergo a 12-week VN intervention in addition to usual medications and nursing home activities, while the control group will continue with their usual medications and activities. Assessments will be performed at baseline, in concomitance with the first VN session, and at 4 and 12 weeks into the intervention.

VN intervention:

The intervention will consist of undergoing a 10-minute VN session twice a week for 12 consecutive weeks. The participants will choose a 360° video from a library of different VN scenarios. The 360° videos within the library will be filmed by the researchers in locations near or in the same region of the participant's nursing homes, and will consist of scenes from various seasons in Norway (spring, summer, fall, winter) and depict popular outdoor recreations such as hiking and cross-country skiing. The VN sessions will be delivered in the participants' room. The playback will be done through a Meta Quest 3 (Reality Labs

, USA). The intervention will be delivered by the researchers in collaboration with caregivers and/or nursing students in practice.

Participants:

Sixty nursing home residents with dementia will be recruited from different nursing homes in Drammen municipality and randomly assigned to the treatment or the control condition. The treatment group will undergo the VN intervention while continuing to receive their usual medications and attending regular activities at their respective nursing homes. The control group will only continue receiving their usual medication and attending regular activities at their respective nursing homes. Inclusion criteria are: being a nursing-home resident with a dementia diagnosis, having normal or corrected-to-normal sight and being able to communicate in Norwegian. Additionally, participants will be excluded if deemed to have poor tolerance to the VN experience (this will be evaluated based on preliminary trials and discussions with caregivers). Written informed consent will be collected for all participants (either directly from the participant or, in case they are not legally competent, their caregivers), after having explained the benefits and risks of participating to them.

Instruments:

Basic demographic data (age and gender) will be recorded. To assess potential long-term effects, the following measures will be collected at baseline, week 4, and week 12 for both the treatment and control groups: Quality of Life in Late-stage Dementia scale, Cornell Scale for Depression in Dementia, Brief Agitation Rating Scale, Clinical Dementia Rating scale, and Use of psychotropic drugs.

ELIGIBILITY:
Inclusion Criteria:

* Nursing-home resident
* Dementia or pre-dementia

Exclusion Criteria:

* Sub-normal sight even when corrected
* Unable to communicate in Norwegian
* Reported or exhibited high intolerance to VN exposure

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Quality of Life in Late-stage Dementia scale | Before the intervention (baseline)
  The Quality of Life in Late-Stage Dementia (QUALID) scale is an observational tool used to assess quality of life in individuals with advanced dementia. It consists of 11 items that evaluate various aspects of well-being, including physical comfort, social interaction, and emotional state. The scale is completed by caregivers or healthcare professionals based on their observations of the individual's behavior and condition. Each item is rated on a 5-point scale, resulting in a total score ranging from 11 to 55, where lower scores indicate better quality of life. The QUALID scale is widely used to assess the impact of interventions and care strategies, helping to ensure comfort and dignity in the final stages of life.
Quality of Life in Late-stage Dementia scale | During the intervention (4 weeks)
  The Quality of Life in Late-Stage Dementia (QUALID) scale is an observational tool used to assess quality of life in individuals with advanced dementia. It consists of 11 items that evaluate various aspects of well-being, including physical comfort, social interaction, and emotional state. The scale is completed by caregivers or healthcare professionals based on their observations of the individual's behavior and condition. Each item is rated on a 5-point scale, resulting in a total score ranging from 11 to 55, where lower scores indicate better quality of life. The QUALID scale is widely used to assess the impact of interventions and care strategies, helping to ensure comfort and dignity in the final stages of life.
Quality of Life in Late-stage Dementia scale | Immediately after the intervention (12 weeks)
  The Quality of Life in Late-Stage Dementia (QUALID) scale is an observational tool used to assess quality of life in individuals with advanced dementia. It consists of 11 items that evaluate various aspects of well-being, including physical comfort, social interaction, and emotional state. The scale is completed by caregivers or healthcare professionals based on their observations of the individual's behavior and condition. Each item is rated on a 5-point scale, resulting in a total score ranging from 11 to 55, where lower scores indicate better quality of life. The QUALID scale is widely used to assess the impact of interventions and care strategies, helping to ensure comfort and dignity in the final stages of life.

SECONDARY OUTCOMES:
Cornell Scale for Depression in Dementia | Before the intervention (baseline)
  The Cornell Scale for Depression in Dementia (CSDD) is a clinician-administered assessment tool developed to evaluate depressive symptoms in individuals with dementia. It combines information from direct interviews with the patient and observations reported by caregivers, allowing for the detection of mood-related symptoms that may not be reliably self-reported due to cognitive impairment. The scale includes 19 items across domains such as mood, behavior, physical signs, and circadian functions. Each item is rated on a 3-point scale (0 = absent, 1 = mild or intermittent, 2 = severe), resulting in a total score ranging from 0 to 38, where higher scores indicate more severe depressive symptoms. The CSDD is commonly used in both clinical and research contexts to identify and monitor depression in individuals with dementia.
Cornell Scale for Depression in Dementia | During the intervention (4 weeks)
  The Cornell Scale for Depression in Dementia (CSDD) is a clinician-administered assessment tool developed to evaluate depressive symptoms in individuals with dementia. It combines information from direct interviews with the patient and observations reported by caregivers, allowing for the detection of mood-related symptoms that may not be reliably self-reported due to cognitive impairment. The scale includes 19 items across domains such as mood, behavior, physical signs, and circadian functions. Each item is rated on a 3-point scale (0 = absent, 1 = mild or intermittent, 2 = severe), resulting in a total score ranging from 0 to 38, where higher scores indicate more severe depressive symptoms. The CSDD is commonly used in both clinical and research contexts to identify and monitor depression in individuals with dementia.
Cornell Scale for Depression in Dementia | Immediately after the intervention (12 weeks)
  The Cornell Scale for Depression in Dementia (CSDD) is a clinician-administered assessment tool developed to evaluate depressive symptoms in individuals with dementia. It combines information from direct interviews with the patient and observations reported by caregivers, allowing for the detection of mood-related symptoms that may not be reliably self-reported due to cognitive impairment. The scale includes 19 items across domains such as mood, behavior, physical signs, and circadian functions. Each item is rated on a 3-point scale (0 = absent, 1 = mild or intermittent, 2 = severe), resulting in a total score ranging from 0 to 38, where higher scores indicate more severe depressive symptoms. The CSDD is commonly used in both clinical and research contexts to identify and monitor depression in individuals with dementia.
Brief Agitation Rating Scale | Before the intervention (baseline)
  The Brief Agitation Rating Scale (BARS) is an observational assessment tool developed to measure the severity of agitation in individuals with cognitive impairments, including dementia. The scale includes 10 items that evaluate behaviors such as restlessness, irritability, verbal aggression, and physical aggression. Each item is rated on a 4-point scale (0 = not present, 1 = mild, 2 = moderate, 3 = severe), resulting in a total score ranging from 0 to 30, where higher scores indicate more severe agitation. The BARS is designed to be brief and practical, enabling quick assessment by caregivers or clinicians in both clinical and research settings.
Brief Agitation Rating Scale | During the intervention (4 weeks)
  The Brief Agitation Rating Scale (BARS) is an observational assessment tool developed to measure the severity of agitation in individuals with cognitive impairments, including dementia. The scale includes 10 items that evaluate behaviors such as restlessness, irritability, verbal aggression, and physical aggression. Each item is rated on a 4-point scale (0 = not present, 1 = mild, 2 = moderate, 3 = severe), resulting in a total score ranging from 0 to 30, where higher scores indicate more severe agitation. The BARS is designed to be brief and practical, enabling quick assessment by caregivers or clinicians in both clinical and research settings.
Brief Agitation Rating Scale | Immediately after the intervention (12 weeks)
  The Brief Agitation Rating Scale (BARS) is an observational assessment tool developed to measure the severity of agitation in individuals with cognitive impairments, including dementia. The scale includes 10 items that evaluate behaviors such as restlessness, irritability, verbal aggression, and physical aggression. Each item is rated on a 4-point scale (0 = not present, 1 = mild, 2 = moderate, 3 = severe), resulting in a total score ranging from 0 to 30, where higher scores indicate more severe agitation. The BARS is designed to be brief and practical, enabling quick assessment by caregivers or clinicians in both clinical and research settings.
Clinical Dementia Rating scale | Before the intervention (baseline)
  The Clinical Dementia Rating (CDR) scale is a widely used clinical tool for assessing the severity of dementia by evaluating both cognitive and functional decline. It examines six domains: memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. Each domain is scored on a 5-point scale, ranging from "no impairment" to "severe impairment". The total CDR score (0, 0.5, 1, 2, or 3) reflects the overall stage of dementia, where higher scores indicate more severe impairment.
Clinical Dementia Rating scale | During the intervention (4 weeks)
  The Clinical Dementia Rating (CDR) scale is a widely used clinical tool for assessing the severity of dementia by evaluating both cognitive and functional decline. It examines six domains: memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. Each domain is scored on a 5-point scale, ranging from "no impairment" to "severe impairment". The total CDR score (0, 0.5, 1, 2, or 3) reflects the overall stage of dementia, where higher scores indicate more severe impairment.
Clinical Dementia Rating scale | Immediately after the intervention (12 weeks)
  The Clinical Dementia Rating (CDR) scale is a widely used clinical tool for assessing the severity of dementia by evaluating both cognitive and functional decline. It examines six domains: memory, orientation, judgment and problem-solving, community affairs, home and hobbies, and personal care. Each domain is scored on a 5-point scale, ranging from "no impairment" to "severe impairment". The total CDR score (0, 0.5, 1, 2, or 3) reflects the overall stage of dementia, where higher scores indicate more severe impairment.
Use of psychotropic drugs | Before the intervention (baseline)
  Use of psychotropic drugs, as reported by nursing staff, including medications for mood disorders, anxiety, depression, and sleep disturbances, are commonly prescribed to manage symptoms in dementia patients. Nursing staff are asked to provide detailed information on the types, dosages, and frequency of psychotropic drugs administered to residents throughout the study period. This measure will help evaluate potential changes in medication usage related to the virtual nature intervention, providing insight into its effects on behavioral and psychological symptoms of dementia.
Use of psychotropic drugs | During the intervention (4 weeks)
  Use of psychotropic drugs, as reported by nursing staff, including medications for mood disorders, anxiety, depression, and sleep disturbances, are commonly prescribed to manage symptoms in dementia patients. Nursing staff are asked to provide detailed information on the types, dosages, and frequency of psychotropic drugs administered to residents throughout the study period. This measure will help evaluate potential changes in medication usage related to the virtual nature intervention, providing insight into its effects on behavioral and psychological symptoms of dementia.
Use of psychotropic drugs | Immediately after the intervention (12 weeks)
  Use of psychotropic drugs, as reported by nursing staff, including medications for mood disorders, anxiety, depression, and sleep disturbances, are commonly prescribed to manage symptoms in dementia patients. Nursing staff are asked to provide detailed information on the types, dosages, and frequency of psychotropic drugs administered to residents throughout the study period. This measure will help evaluate potential changes in medication usage related to the virtual nature intervention, providing insight into its effects on behavioral and psychological symptoms of dementia.

OTHER OUTCOMES:
Age | Before the intervention (baseline)
  Participant's age, as reported by the nursing-home staff
Gender | Before the intervention (baseline)
  Participant's gender, as reported by the nursing-home staff

CONTACTS AND LOCATIONS:
Overall Officials: Giovanna Calogiuri, Principal Investigator — University of South-Eastern Norway

REFERENCES:
- [Background] Morris JC. The Clinical Dementia Rating (CDR): current version and scoring rules. Neurology. 1993 Nov;43(11):2412-4. doi: 10.1212/wnl.43.11.2412-a. No abstract available. PMID 8232972
- [Background] Finkel SI, Lyons JS, Anderson RL. A brief agitation rating scale (BARS) for nursing home elderly. J Am Geriatr Soc. 1993 Jan;41(1):50-2. doi: 10.1111/j.1532-5415.1993.tb05948.x. PMID 8418123
- [Background] Alexopoulos GS, Abrams RC, Young RC, Shamoian CA. Cornell Scale for Depression in Dementia. Biol Psychiatry. 1988 Feb 1;23(3):271-84. doi: 10.1016/0006-3223(88)90038-8. PMID 3337862
- [Background] Roen I, Selbaek G, Kirkevold O, Engedal K, Lerdal A, Bergh S. The Reliability and Validity of the Norwegian Version of the Quality of Life in Late-Stage Dementia Scale. Dement Geriatr Cogn Disord. 2015;40(3-4):233-42. doi: 10.1159/000437093. Epub 2015 Jul 28. PMID 26227299
- See also: Poster presented at the Norwegian Public Health conference, October 24-25, 2024, Tønsberg, Norway — https://folkehelsekonferansen.no/dokumenter/F-FHK24-Giovanna-Calogiuri.pdf